CLINICAL TRIAL: NCT01367457
Title: Inhibitor - Estudio Retrospectivo De Casos Clinicos De Pacientes Con Carcinoma De Celulas Renales Y Con Linforma De Celulas Del Manto Tratados Con Temsirolimus
Brief Title: INHIBITOR: Retrospective Study Of Patients With Renal Cell Carcinoma And Mantle Cell Lymphoma Treated With Temsirolimus
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B1771017; INHIBITOR (Other: Alias Study Number)
Record Dates: First submitted 2011-06-03; First posted 2011-06-07 (Estimated); Results first posted 2016-04-27 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2016-03

CONDITIONS: Carcinoma, Renal Cell; Lymphoma, Mantle-Cell
MeSH Terms: conditions — Carcinoma, Renal Cell; Lymphoma, Mantle-Cell | interventions — temsirolimus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients that received treatment with Temsirolimus: Patients with Renal Cell Carcinoma or Mantle Cell Lymphoma that have been treated with Temsirolimus as per clinical practice.
  Interventions: Other: Temsirolimus (Non-Interventional Study)

INTERVENTIONS:
Other: Temsirolimus (Non-Interventional Study) — There is not any intervention in this study.

SUMMARY:
The principal objective of the study is to evaluate the efficacy and safety of temsirolimus use in patients with Renal Cell Carcinoma and Mantle Cell Lymphoma.

DETAILED DESCRIPTION:
There is not sampling method

ELIGIBILITY:
Inclusion Criteria:

Patients with Renal Cell Carcinoma or Mantle Cell Lymphoma that have been treated with Temsirolimus as per clinical practice.

Exclusion Criteria:

Patients that do not have a minimum (pre-specified) of data in their clinical record.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Renal Cell Carcinoma or Mantle Cell Lymphoma that have been treated with Temsirolimus as per clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 243 (Actual)
Dates: Start 2011-01; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (16):
- Spain (16):
  - Complexo Hospitalario Universitario A Coruña, A Coruña, A Coruña
  - Hospital de La Santa Creu I Sant Pau, Barcelona, Barcelona
  - Hospital Vall D'Hebron, Barcelona, Barcelona
  - Hospital del Mar, Barcelona, Barcelona
  - Hospital de Cabueñes, Cabueñes, Gijon
  - Complexo Hospitalario Universitario A Coruña. Hospital Teresa Herrera, A Coruña, La Coruña
  - Hospital Clinico Universitario, Santiago de Compostela, La Coruña
  - Complejo Hospitalario Materno-Infantil Insular de Las Palmas, Las Palmas de Gran Canaria, Las Palmas
  - Hospital General Universitario Gregorio Marañon, Madrid, Madrid
  - Hospital Universitario La Paz, Madrid, Madrid
  - Hospital de Madrid Norte - Sanchinarro, Madrid, Madrid
  - Hospital de Navarra, Pamplona, Navarre
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Provincial de Castellon, Castellon, Valencia
  - Complejo AAsistencial de Avilla, Ávila
  - MD Anderson Cancer Center, Madrid

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1771017&StudyName=INHIBITOR%3A%20Retrospective%20Study%20Of%20Patients%20With%20Renal%20Cell%20Carcinoma%20And%20Mantle%20Cell%20Lymphoma%20Treated%20With%20Temsirolimus

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 243 participants were enrolled in the study, out of which 242 participants received treatment in reporting group "RCC: Temsirolimus", "MCL: Temsirolimus" or "MCL: Temsirolimus + Rituximab"
Groups:
- RCC: Temsirolimus: Participants diagnosed with Renal Cell Carcinoma (RCC) who received treatment with Temsirolimus as per standard clinical practice and received at least 1 dose of Temsirolimus were included in this non-interventional study.
- MCL: Temsirolimus: Participants diagnosed with Mantle Cell Lymphoma (MCL) who received treatment with Temsirolimus as per standard clinical practice and received at least 1 dose of Temsirolimus as monotherapy were included in this non-interventional study.
- MCL: Temsirolimus + Rituximab: Participants diagnosed with MCL who received treatment with Temsirolimus as per standard clinical practice and received at least 1 dose of Temsirolimus as combination therapy with Rituximab.
Period: Overall Study
Arm/Group | RCC: Temsirolimus | MCL: Temsirolimus | MCL: Temsirolimus + Rituximab
Started | 193 | 23 | 26
Completed | 5 | 23 | 26
Not Completed | 188 | 0 | 0
Not completed — Death | 2 | 0 | 0
Not completed — Investigator's decision | 2 | 0 | 0
Not completed — Clinical decline (CD) | 2 | 0 | 0
Not completed — Progression and death | 8 | 0 | 0
Not completed — Toxicity | 16 | 0 | 0
Not completed — Progression | 137 | 0 | 0
Not completed — Patient asks for rest + slow progression | 1 | 0 | 0
Not completed — Investigator's opinion, stable disease | 1 | 0 | 0
Not completed — Bleeding from cavernous haemangioma | 1 | 0 | 0
Not completed — 3 yr Temsirolimus treatment (no disease) | 1 | 0 | 0
Not completed — low grade toxicities + stable disease | 1 | 0 | 0
Not completed — Choledocolithiasis and pancreatitis | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — CD, associated leukaemia | 1 | 0 | 0
Not completed — Uncontrolled pain | 1 | 0 | 0
Not completed — Overall status worsens to grade 4 | 1 | 0 | 0
Not completed — Stabilisation + frequent infections | 1 | 0 | 0
Not completed — No clinical benefit | 1 | 0 | 0
Not completed — Intestinal obstruction with necrosis | 1 | 0 | 0
Not completed — Overall decline | 1 | 0 | 0
Not completed — Rejection of treatment | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Death from septic shock | 1 | 0 | 0
Not completed — CD, Suspected disease progression (DP) | 1 | 0 | 0
Not completed — Patient's Wish | 1 | 0 | 0
Not completed — Palliative. Overall decline | 1 | 0 | 0
Not completed — Suspected DP/suspected active infection | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline population included all participants with RCC or MCL who received atleast 1 dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | RCC: Temsirolimus | MCL: Temsirolimus | MCL: Temsirolimus + Rituximab | Total
Number analyzed (Participants) | 193 | 23 | 26 | 242
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.27 (11.14) | 70.56 (11.07) | 72.34 (7.11) | 66.54 (11.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 3 | 3 | 63
  Male | 136 | 20 | 23 | 179

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival: interval between start of treatment to first day when progressive disease (PD) was evaluated according to Response Evaluation Criteria in Solid Tumors (RECIST) for participants with RCC and Cheson criteria for participants with MCL, or death due to any cause. RECIST criteria: at least 20% increase in sum of diameters of target lesions, taking as reference the smallest sum. In addition to relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 millimeter (mm). Appearance of one or more new lesions also considered progression. Cheson criteria: appearance of any new sites of lymphoma OR at least 50% increase in product of longest perpendicular dimensions of any previously identified lymph node mass (LNM) OR at least 50% increase in longest dimension of any previously identified LNM greater than 1 cm in longest transverse dimension OR at least 50% increase in size of any previously involved site of lymphoma.
Time Frame: From initiation of treatment up to disease progression (up to 80 months)
Population: Evaluable population included all participants with RCC or MCL who received atleast 1 dose of study treatment.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- MCC: Temsirolimus + Rituximab: Participants diagnosed with MCL who received treatment with Temsirolimus as per standard clinical practice and received at least 1 dose of Temsirolimus as combination therapy with Rituximab.
Arm/Group | RCC: Temsirolimus | MCL: Temsirolimus | MCC: Temsirolimus + Rituximab
Number analyzed (Participants) | 193 | 23 | 26
months | 4.04 [3.03 to 5.05] | 7.467 [4.171 to 10.763] | 13.233 [3.306 to 23.161]

2. Primary Outcome: Percentage of Participants With Objective Response
Description: Objective response: percentage of participants who achieved complete remission (CR) or partial response (PR). RECIST criteria was used for participants with RCC and Cheson criteria for participants with MCL. RECIST criteria (CR: disappearance of all target lesions, any pathological lymph nodes(target or non-target) reduced in short axis to <10 mm, PR: at least 30% decrease in sum of diameters of target lesions). Cheson criteria (CR: all lymph node masses regressed to normal size, each lymph node mass that was >1.5 cm in longest transverse dimension regressed to <=1.5 cm, lymph node mass that was 1.1-1.5 cm regressed to <=1 cm, complete disappearance of all radiographic evidence of disease, PR: at least 50% decrease in sum of products of the longest perpendicular dimensions of the previously identified dominant lymph node masses, no increase in size of other lymph nodes.)
Time Frame: From initiation of treatment up to disease progression (up to 80 months)
Population: Evaluable population included all participants with RCC or MCL who received atleast 1 dose of study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | RCC: Temsirolimus | MCL: Temsirolimus | MCC: Temsirolimus + Rituximab
Number analyzed (Participants) | 193 | 23 | 26
percentage of participants
  CR | 0.5 | 34.8 | 30.8
  PR | 14.3 | 17.4 | 50.0
  SD | 46.6 | 26.1 | 7.7
  DP | 38.6 | 21.7 | 11.5

3. Primary Outcome: Duration of Response (DOR)
Description: Duration of response (DOR) was defined as the interval from the date the response was documented to the first date that progression of disease (PD) was observed in participants with PR or CR. RECIST criteria was used for participants with RCC and Cheson criteria for participants with MCL. PD, CR and PR are defined in primary outcome 1 and 2.
Time Frame: From initiation of treatment up to disease progression (up to 80 months)
Population: Evaluable population included all participants with RCC or MCL who received atleast 1 dose of study treatment. Here, number of participants analyzed signifies those participants who were evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | RCC: Temsirolimus | MCL: Temsirolimus | MCC: Temsirolimus + Rituximab
Number analyzed (Participants) | 28 | 12 | 20
months | 13.21 [8.55 to 17.87] | 7.28 [4.23 to 9.85] | 8.82 [6.42 to 13.16]

4. Primary Outcome: Overall Survival (OS)
Description: Overall survival (OS) was defined as the interval from the day of the start of the treatment to death, or censored to the last date when the participant was identified to be alive.
Time Frame: From initiation of treatment untill death (up to 80 months)
Population: Evaluable population included all participants with RCC or MCL who received atleast 1 dose of study treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | RCC: Temsirolimus | MCL: Temsirolimus | MCC: Temsirolimus + Rituximab
Number analyzed (Participants) | 193 | 23 | 26
months | 10.81 [8.20 to 13.42] | 19.233 [3.052 to 35.415] | 18.667 [NA to NA] — The last event had happened when function survival reached the median value.

5. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent events were between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state. AEs included both SAEs and non-serious adverse events (Non-SAEs).
Time Frame: Baseline to the 28 calendar days after the last administration of study drug (upto 80 months)
Population: Safety population included all participants with RCC or MCL who received atleast 1 dose of study treatment.
Measure: Number; unit: participants
Arm/Group | RCC: Temsirolimus | MCL: Temsirolimus | MCC: Temsirolimus + Rituximab
Number analyzed (Participants) | 193 | 23 | 26
participants
  AEs | 145 | 19 | 16
  SAEs | 18 | 3 | 7

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant or one participant may have experienced both a serious and non-serious event during the study.
Arm/Group | RCC: Temsirolimus | MCL: Temsirolimus | MCL: Temsirolimus + Rituximab
Serious Adverse Events (participants affected / at risk) | 18/193 | 3/23 | 7/26
Other Adverse Events (participants affected / at risk) | 142/193 | 18/23 | 14/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RCC: Temsirolimus (N=193) | MCL: Temsirolimus (N=23) | MCL: Temsirolimus + Rituximab (N=26)
Death (General disorders) | 1 | 0 | 0
Disease progression (General disorders) | 2 | 0 | 0
Malaise (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal toxicity (Gastrointestinal disorders) | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Haemangioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Coma (Nervous system disorders) | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0 | 0
Others (General disorders) | 1 | 0 | 2 — No coding was available in MedDRA dictionary for this event
Aspergillus infection (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RCC: Temsirolimus (N=193) | MCL: Temsirolimus (N=23) | MCL: Temsirolimus + Rituximab (N=26)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 19 | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 23 | 3 | 2
Hyperlipidaemia (Metabolism and nutrition disorders) | 11 | 2 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 5 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 13 | 1 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypertriglyceridemia (Metabolism and nutrition disorders) | 8 | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 58 | 4 | 3
Leukopenia (Blood and lymphatic system disorders) | 2 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 4 | 1 | 3
Bone marrow toxicity (Blood and lymphatic system disorders) | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 11 | 12 | 5
Stomatitis (Gastrointestinal disorders) | 41 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Chronic gastritis (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 5 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 13 | 3 | 4
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 6 | 1 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 9 | 0 | 0
Asthenia (General disorders) | 43 | 4 | 1
Malaise (General disorders) | 1 | 0 | 0
Mucosal inflammation (General disorders) | 3 | 2 | 1
Oedema (General disorders) | 3 | 1 | 0
Oedema peripheral (General disorders) | 4 | 0 | 0
Pain (General disorders) | 3 | 0 | 0
Pyrexia (General disorders) | 6 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin toxicity (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dermal toxicity (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Nail toxicity (Skin and subcutaneous tissue disorders) | 5 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 0 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 26 | 2 | 3
Skin mass (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 17 | 2 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Tonsillar disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 2 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0
Blood creatinine increased (Investigations) | 6 | 0 | 0
Transaminases increased (Investigations) | 1 | 0 | 0
Polyuria (Renal and urinary disorders) | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 7 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 1
Dysgeusia (Nervous system disorders) | 4 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 0
Neuralgia (Nervous system disorders) | 1 | 0 | 0
Sciatica (Nervous system disorders) | 1 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 1
Gastrointestinal candidiasis (Infections and infestations) | 0 | 0 | 1
Gingivitis (Infections and infestations) | 2 | 0 | 0
Infection (Infections and infestations) | 2 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 2
Oral candidiasis (Infections and infestations) | 0 | 0 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 2
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 2
Infusion related reaction (Injury, poisoning and procedural complications) | 2 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 1 | 0
Eyelids pruritus (Eye disorders) | 1 | 0 | 0
Visual acuity reduced (Eye disorders) | 0 | 0 | 1
Cholestasis (Hepatobiliary disorders) | 0 | 0 | 1
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0
Aortic aneurysm (Vascular disorders) | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0
Embolism (Vascular disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1
Thrombophlebitis (Vascular disorders) | 0 | 0 | 1
Others (General disorders) | 3 | 1 | 2 — No coding was available in MedDRA dictionary for this event
Herpes zoster (Infections and infestations) | 2 | 0 | 0
Deafness (Ear and labyrinth disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.